CLINICAL TRIAL: NCT06545448
Title: Appropriateness of Angioplasty in Patients With Chronic Coronary Syndromes in a Cardiology Reference Hospital - The RIGHT-PCI Study
Brief Title: Appropriateness of Angioplasty in Patients With Chronic Coronary Syndromes
Acronym: RIGHT-PCI
Status: Recruiting | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Sponsor
Other Study IDs: 70150723.8.0000.0068
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Coronary Artery Disease; Angina Pectoris
Keywords: Coronary artery disease; Angina pectoris; Angioplasty; Appropriateness; Prognosis; Treatment
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris | interventions — Percutaneous Coronary Intervention; Angioplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing elective PCI: Patients undergoing elective PCI for chronic coronary syndrome in a tertiary hospital in a single center in Brazil between 2017-2020.
  Interventions: Procedure: Percutaneous Coronary Intervention (PCI)

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention (PCI) — A percutaneous coronary intervention (PCI) is a minimally invasive procedure to open blocked coronary (heart) arteries. An older name for PCI is coronary angioplasty with stenting or angioplasty for short.
  Other Names: Angioplasty

SUMMARY:
Percutaneous coronary intervention (PCI) has dramatically changed the treatment of obstructive coronary artery disease patients. PCI is indicated in patients with chronic coronary syndrome (CCS) symptoms unresponsive to optimized medical therapy. The American College of Cardiology Foundation and partners developed in 2009 - and updated them in May 2017 - the appropriateness criteria for PCI to support the rational use of PCI in chronic patients and to provide patients with high-quality cardiovascular care. Since then, these criteria have been applied to guide physicians and serve as metrics of the quality of care based on the best available scientific evidence. Countries like the United States and Japan already have robust studies on the topic with important repercussions on clinical practice. In Brazil, to date, there are no studies on the adequacy of PCIs in patients with CCS.

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) has dramatically changed the treatment of obstructive coronary artery disease patients. PCI is indicated in patients with chronic coronary syndrome (CCS) symptoms unresponsive to optimized medical therapy. The American College of Cardiology Foundation and partners developed in 2009 - and updated them in May 2017 - the appropriateness criteria for PCI to support the rational use of PCI in chronic patients and to provide patients with high-quality cardiovascular care. Since then, these criteria have been applied to guide physicians and serve as metrics of the quality of care based on the best available scientific evidence. Countries like the United States and Japan already have robust studies on the topic with important repercussions on clinical practice. In Brazil, to date, there are no studies on the adequacy of PCIs in patients with CCS.

The primary goal of the RIGHT-PCI study is to determine the rate of PCI indications categorized as appropriate, possibly appropriate, or rarely appropriate in patients with CCS undergoing elective PCI based on criteria established in medical literature at a Cardiology reference university hospital. To achieve this objective, we plan to analyze approximately 2,500 consecutive angioplasties performed between 2017 and 2020.

ELIGIBILITY:
Inclusion Criteria:

* All patients within the age range who underwent elective PCI defined as a procedure indicated in an outpatient scenario or an inpatient in a non-acute setting when the Heart Team was called to evaluate the patient and agreed with the indication for PCI

Exclusion Criteria:

* History of acute coronary syndrome < 30 days of the referral for PCI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients within the age range who underwent elective PCI indicated their own physicians. This procedure was defined as an outpatient scenario or an inpatient in a non-acute setting when the Heart Team was called to evaluate the patient and agreed with the indication for PCI.
Sampling Method: Non-Probability Sample
Enrollment: 1875 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine the rates of elective PCI classified as appropriate, possibly appropriate, or rarely appropriate. | Immediately following the procedure
  Determine the rates of elective PCI classified as appropriate, possibly appropriate, or rarely appropriate based on the Appropriateness Criteria proposed by the ACC / AHA in 2017.

SECONDARY OUTCOMES:
Incidence of the composite endpoint of all-cause mortality and non-fatal cardiovascular events (myocardial infarction, periprocedural stroke, or the need for new revascularization) | 12 months after the procedure index
  Incidence of the composite endpoint of all-cause mortality and non-fatal cardiovascular events (myocardial infarction based on the 4th Universal Definition of MI, periprocedural stroke occurring during the hospitalization index, or the need for new revascularization either by CABG or PCI)
Incidence of persistent or recurrent post-PCI angina or new onset/worsening heart failure | 12 months after the procedure index
  Incidence of persistent or recurrent post-PCI angina or new onset/worsening heart failure both clinically manifest

OTHER OUTCOMES:
Clinical and sociodemographic predictors of rarely appropriate elective PCI | Immediately following the procedure
  Clinical and sociodemographic predictors of rarely appropriate elective PCI

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Institute (InCor-HCFMUSP), São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
There is no formal plan yet, but our team will consider any suggestions for a joint study.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 5 years from the first publication
Access Criteria: By e-mail only